CLINICAL TRIAL: NCT04012684
Title: Using Repetitive Transcranial Magnetic Stimulation to Improve the Auditory Mismatch Negativity Deficits of Schizophrenia: a Randomized, Double-blinded, Sham-controlled Clinical Trial
Brief Title: rTMS on Mismatch Negativity of Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201807026RINB
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia; Mismatch Negativity
Keywords: Repetitive transcranial stimulation; Inferior frontal gyrus
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS: left first (Experimental): One-session rTMS is applied to left IFG. Pre-stimulation and post-stimulation MMN is recorded and compared. After at least two weeks, one-session rTMS is applied to right IFG. Pre-stimulation and post-stimulation MMN is recorded and compared as well.
  Interventions: Device: Transcranial magnetic stimulation
- rTMS: right first (Experimental): One-session rTMS is applied to right IFG. Pre-stimulation and post-stimulation MMN is recorded and compared. After at least two weeks, one-session rTMS is applied to left IFG. Pre-stimulation and post-stimulation MMN is recorded and compared as well.
  After at least two weeks, stimulations of the same parameters are given over left IFG. Pre-stimulation and post-stimulation MMN is recorded and compared as well.
  Interventions: Device: Transcranial magnetic stimulation
- Sham: left first (Sham Comparator): One-session sham stimulation is applied to left IFG. Pre-stimulation and post-stimulation MMN is recorded and compared. After at least two weeks, one-session sham stimulation is applied to right IFG. Pre-stimulation and post-stimulation MMN is recorded and compared as well.
  Interventions: Device: Sham
- Sham: right first (Sham Comparator): One-session sham stimulation is applied to right IFG. Pre-stimulation and post-stimulation MMN is recorded and compared. After at least two weeks, one-session sham stimulation is applied to left IFG. Pre-stimulation and post-stimulation MMN is recorded and compared as well.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial magnetic stimulation — For one-session rTMS, 50 trains of stimulation are given. Each train is consisted of 4-second 10 Hz, 100% resting motor threshold TMS pulses. The inter-train interval is 26 seconds.
  Arms: rTMS: left first; rTMS: right first
Device: Sham — For one-session sham stimulation, 50 trains of stimulation are given. Each train is consisted of 4-second 10 Hz sham pulses. The inter-train interval is 26 seconds.
  Arms: Sham: left first; Sham: right first

SUMMARY:
Auditory mismatch negativity deficit is a robust neurophysiological biomarker of schizophrenia. Repetitive transcranial magnetic stimulation (rTMS) is a neuromodulation method and can be used to modulate excitability of specific brain cortical region. We hypothesize that MMN deficit of schizophrenia is related to inferior frontal gyrus (IFG) hypofunction, and this deficit can be improved by using rTMS to enhance IFG function.

It is a randomized, double-blinded, sham-controlled clinical trial. Forty-eight schizophrenia patients with MMN deficits (mean amplitude at FCz > -0.7 ㎶) will be recruited and then randomized at a 1:1 ratio to rTMS group and sham-stimulation group. Subjects in rTMS group will receive high frequency rTMS over IFG, while in the other group subjects will receive sham stimulation at IFG. Frameless stereotaxy navigation will be used to guide the rTMS coil to IFG. The primary outcome is the change of MMN mean amplitude at FCz after stimulation. We hypothesize that the change of MMN mean amplitude is significantly larger in rTMS group than in sham-stimulation group. Their cognitive function and clinical condition will be evaluated carefully before and after experiments.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision
* mean amplitude of MMN at FCz greater than -0.7 ㎶
* moderate or milder disease severity (scoring 4 or below according to clinical global rating scale)

Exclusion Criteria:

* unwillingness or inability to cooperate with the experiments
* with mental retardation, epilepsy, or other major brain pathology (e.g. cerebrovascular accidents or major head injury)
* with alcohol or other illicit substance abuse
* with major debilitating systemic diseases or difficulties in ambulation
* with hearing impairments as screened by audiometry over 500 Hz, 1000 Hz and 6000 Hz
* with pacemaker, intra-ocular metal foreign body, intracerebral vessel clip, artificial cardiac valve, electronic implant in the body, claustrophobia, or previous surgery involving the brain
* being pregnant or to be pregnant during the clinical trial. A pre-TMS evaluation scale will be applied to ensure the safety

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Mismatch negativity (MMN) | 1 day
  Mismatch negativity is recorded by electroencephalography and elicited by auditory oddball paradigm in which tone duration deviants are used. MMN is the mean amplitude between 135 and 205 milliseconds after auditory stimuli recorded by electrode FCz.

SECONDARY OUTCOMES:
Continuous performance test (CPT) | 1 day
  The undegraded 1-9 task and the 25% degraded 1-9 task are used. Sensitivity indices indicating the ability to discriminate target from non-target trials are calculated (d' for undegraded CPT and md' for degraded CPT).
Wisconsin Card Sorting Test (WCST) | 1 day
  Four indices of WCST are derived: perseverative errors, categories achieved, trials to complete first category, and conceptual level response.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan